CLINICAL TRIAL: NCT02867150
Title: A Retrospective Analysis of the Effects of Red Light Therapy on Body Contouring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ward Photonics LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MLS-1510
Record Dates: First submitted 2016-01-03; First posted 2016-08-15 (Estimated); Results first posted 2017-06-23 (Actual); Last update posted 2017-06-23 (Actual); Status verified 2017-06

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Active Device (Experimental): Active Device: Ward Photonics Photonica Professional Red light therapy system Intervention: Device: Ward Photonics Photonica Professional
  Interventions: Device: Ward Photonics Photonica Professional

INTERVENTIONS:
Device: Ward Photonics Photonica Professional — Active Device: Ward Photonics, Photonica Professional Red light therapy system
  UltraSlim Cold Light® is the name of a patented treatment regimen using the Photonica Professional device for fat removal using LED red light therapy.

SUMMARY:
The purpose of this study is to determine whether red light therapy using LED 635nm red light for body contouring of the waist, hips and thighs is as effective as red light therapy using Laser 635nm red light.

DETAILED DESCRIPTION:
Red light laser therapy using 635nm red light laser technology has previously been shown to cause lipolysis in subcutaneous fat as a non-surgical method to promote weight loss and body contouring. This study hypothesizes that red LED light therapy using 635nm red light LED (light emitting diode) technology produces similar results to the laser device (red LASER 635nm) when performed using a specified treatment protocol.

Furthermore, it is hypothesized that the UltraSlim Cold Light therapy program achieves the results after a single 32-minute treatment. The predicate 635nm laser device (Zerona by Erchonia) achieves its results after six treatments combined with a diet and exercise regimen.

UltraSlim Cold Light® is a patented process using the Photonica Professional device for fat removal using LED red light therapy. This multi-site study reviews results from 58 randomly selected patients after a single treatment using the Photonica Professional device (i.e. UltraSlim Cold Light®).

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older.
* Male or female.
* Generally good health.

Exclusion Criteria:

* Pregnancy.
* Active cancer within the past year.
* Diminished ability to void waste (liver or kidneys).
* Photosensitive condition or medication.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2015-10; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Terry J Ward, M.H.A., Principal Investigator — Managing Director

IPD SHARING:
Plan to Share IPD: No
No current plan to share data.

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Device: Active Device: Ward Photonics Photonica Professional Red light therapy system Intervention: Device: Ward Photonics Photonica Professional
  Ward Photonics Photonica Professional: Active Device: Ward Photonics, Photonica Professional Red light therapy system
  UltraSlim Cold Light® is the name of a patented treatment regimen using the Photonica Professional device for fat removal using LED red light therapy.
Period: Overall Study
Arm/Group | Active Device
Started | 58
Completed | 58
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Active Device
Number analyzed (Participants) | 58
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 54
  >=65 years | 3
Age, Continuous [Mean (Full Range); unit: Years] | 43.3 [18 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46
  Male | 12
Region of Enrollment [Number; unit: participants] — Multi-site U.S. Study
  participants
    United States | 58

OUTCOME MEASURES:

1. Primary Outcome: Fat Reduction in Treatment Zone as Measured in Inches Lost
Description: Circumferential measurement of thighs, hips and waist before and after treatment.
Time Frame: Single 32-minute treatment session
Measure: Mean (Full Range); unit: inch
Arm/Group | Active Device
Number analyzed (Participants) | 58
inch | 3.5 [1.625 to 10]

ADVERSE EVENTS:
Time Frame: 6 MONTHS
Description: No observations of any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research.
  Types of adverse events monitored: "All-Cause Mortality," "Serious," and "Other (Not Including Serious)" Adverse Events.
Arm/Group | Active Device
Serious Adverse Events (participants affected / at risk) | 0/58
Other Adverse Events (participants affected / at risk) | 0/58

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No